CLINICAL TRIAL: NCT02740517
Title: Reassure Respiration Rate Device: Home User Study
Brief Title: Usability Evaluation - Reassure Respiration Rate Device: Home User Study
Status: Completed | Type: Observational
Sponsor: ResMed (Industry)
Responsible Party: Sponsor
Other Study IDs: D22105-115
Record Dates: First submitted 2016-04-12; First posted 2016-04-15 (Estimated); Results first posted 2021-05-07 (Actual); Last update posted 2021-05-07 (Actual); Status verified 2021-04

CONDITIONS: Ease of Use

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- HUT1: First phase of the home user trial. 19 users, 12 who were part of a couple and 7 who were single.
- HUT2: Second phase of home user trial, testing improvements to the device user interface as a result of the experience from HUT1. Total 11 users.
  Main change to device was a simpler set of displays and button-sequence on a 24 hour period.
- HUT3: Third phase of home user trial, testing the final improvements to the device. A total of 18 users, 16 of which who were part of a couple and 2 who were single.
  Main change was the introduction of a scheduled recording option, making the device totally automatic in routine use.

SUMMARY:
This is a usability evaluation of the Reassure device. The device is a non-contact device which passively monitors breathing.

The purpose of this usability evaluation is to understand any issues that the intended user population have while using the device unsupervised in the home and to determine if the device can collect data that is of sufficient quality to be successfully analysed for respiration rate.

DETAILED DESCRIPTION:
The aim of the set of Reassure Home User Trials is to understand any usability issues that users have while using the Reassure non contact monitor in their home environment.

Other objectives:

* To gather useful feedback on the user interface and suggestions for its improvement.
* To gather information on the device stability in the more variable conditions of the home user environment.
* To gather data in order to demonstrate compliance with IEC62366, and thus IEC60601-1

The users had the device for a minimum of 10 nights, to confirm if the device could be used for an extended period and the likely compliance rates of users

ELIGIBILITY:
Inclusion Criteria:

* volunteer, no previous exposure to the device

Exclusion Criteria:

* restless leg syndrome or other conditions giving to uncontrolled movements whilst asleep

Ages: 30 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Up to 60 volunteers, all naïve to the device. The majority of the volunteers to be >65 years old, to represent the likely user profile: person with a set of chronic diseases, and not necessarily technically adept
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2014-10; Primary Completion 2015-11 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Phillips, MA, MSc, Principal Investigator — ResMed Sensor Technologies Ltd

IPD SHARING:
Plan to Share IPD: No
Trial to validate the user features of the new medical device. Trial registered with ClinicalTrials.gov only because it involves human volunteers. No plans to publish

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Devices used in the subjects' own homes to monitor their respiration rates whilst asleep in their own beds. Subjects all naïve to the device. A mix of couples and single subjects used. The subjects are predominately senior citizens to replicate the most likely user of the device
Groups:
- Home User Trial Phase 1 (HUT1): First phase of the home user trial.
- Home User Trial Phase 2 (HUT2): Second phase of home user trial, testing improvements to the device user interface as a result of the experience from HUT1.
- Home User Trial Phase 3 (HUT3): Third phase of home user trial, testing the final improvements to the device.
Period: Overall Study
Arm/Group | Home User Trial Phase 1 (HUT1) | Home User Trial Phase 2 (HUT2) | Home User Trial Phase 3 (HUT3)
Started | 19 | 11 | 18
Completed | 19 | 11 | 18
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Home User Trial Phase 1 (HUT1) | Home User Trial Phase 2 (HUT2) | Home User Trial Phase 3 (HUT3) | Total
Number analyzed (Participants) | 19 | 11 | 18 | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 0 | 15 | 19
  >=65 years | 15 | 11 | 3 | 29
Sex/Gender, Customized [Number; unit: participants] | 19 | 11 | 18 | 48
Region of Enrollment [Number; unit: participants]
  Ireland | 19 | 11 | 18 | 48
Part of a Couple [Count of Participants; unit: Participants] | 11 | 11 | 16 | 38
Single [Count of Participants; unit: Participants] | 7 | 0 | 2 | 9

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Nights' Data That Were Successfully Recorded
Description: The definitions utilised to determine the patient's success or otherwise at making a recording of their sleep respiration data are:
  • That 67% of the duration of the recording has to be of sufficient quality for the respiration rate algorithms to be able to discern a respiration rate.
  AND
  • The duration of analysable data is to be at least 2 hours.
Time Frame: At least 10 nights
Measure: Number; unit: percentage of nights' data
Arm/Group | Home User Trial Phase 1 (HUT1) | Home User Trial Phase 2 (HUT2) | Home User Trial Phase 3 (HUT3)
Number analyzed (Participants) | 19 | 11 | 18
percentage of nights' data | 79 | 86 | 100

2. Secondary Outcome: Percentage of Recordings With Successful First Time Transmission
Description: Percentage of the recordings that were successfully transmitted from the home location to the central database on the day of the recording
Time Frame: For at least 10 nights of recordings
Measure: Number; unit: percentage of first time transmissions
Arm/Group | Home User Trial Phase 1 (HUT1) | Home User Trial Phase 2 (HUT2) | Home User Trial Phase 3 (HUT3)
Number analyzed (Participants) | 19 | 11 | 18
percentage of first time transmissions | 49 | 76.7 | 96.7

ADVERSE EVENTS:
Time Frame: 10 days during which the device was being used in the home environment
Arm/Group | Home User Trial Phase 1 (HUT1) | Home User Trial Phase 2 (HUT2) | Home User Trial Phase 3 (HUT3)
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/11 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/11 | 0/18
Other Adverse Events (participants affected / at risk) | 0/19 | 0/11 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes